CLINICAL TRIAL: NCT00945490
Title: Phase III Multicenter Prospective Randomized Parallel-Group Placebo-Controlled Double Blind Clinical Evaluation of NX-1207 for the Treatment of BPH NX02-0018
Brief Title: Clinical Evaluation of NX-1207 for the Treatment of Benign Prostatic Hyperplasia (BPH) NX02-0018
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nymox Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NX02-0018
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
Keywords: Benign prostatic hyperplasia; BPH; Enlarged prostate
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — fexapotide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NX-1207 (Experimental)
  Interventions: Drug: NX-1207
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NX-1207 — Single intraprostatic injection of 2.5 mg NX-1207
  Arms: NX-1207
Drug: Placebo — Single intraprostatic injection of placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of a 2.5 mg dose of NX-1207 for the treatment of BPH (benign prostatic hyperplasia) as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent prior to enrolment in the study
2. AUASI ≥ 15
3. Prostate Volume ≥ 30 mL ≤ 70 mL
4. Qmax < 15 mL/sec based on a minimum void of 125 mL
5. Agree not to use any other approved or experimental BPH or OAB medication anytime during the study

Exclusion Criteria:

1. History of illness or condition that may interfere with study or endanger subject
2. Use of prescribed medications that may interfere with study or endanger subject
3. Presence of a median lobe of the prostate
4. Previous surgery or MIST for treatment of BPH
5. Post-void residual urine volume > 200 mL
6. PSA ≥ 10 ng/mL; prostate cancer must be ruled out (negative biopsy) for PSA ≥ 4 ng/mL
7. Participation in a study of any investigational drug or device within the previous 90 days
8. Prostate cancer

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2009-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
American Urological Association Symptom Index (AUASI) | 365 days

SECONDARY OUTCOMES:
American Urological Association Symptom Index (AUASI) | 90 days
American Urological Association Symptom Index (AUASI) | 180 days
American Urological Association Symptom Index (AUASI) | 270 days
Peak urine flow rate (Qmax) | 365 days
Peak urine flow rate (Qmax) | 90 days
Peak urine flow rate (Qmax) | 180 days

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Laguna Hills, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., San Diego, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Tarzana, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Torrance, California
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Denver, Colorado
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Englewood, Colorado
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Aventura, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Ocala, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Orlando, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Sarasota, Florida
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Meridian, Idaho
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Annapolis, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Baltimore, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Glen Burnie, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Towson, Maryland
  - For information concerning this clinical site, please contact Nymox at 800-936-9669, Grand Rapids, Michigan
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Sartell, Minnesota
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Southaven, Mississippi
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Las Vegas, Nevada
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Brick, New Jersey
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Albuquerque, New Mexico
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Albany, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Garden City, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., New York, New York
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Bismarck, North Dakota
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Oklahoma City, Oklahoma
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Bryn Mawr, Pennsylvania
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Sewickley, Pennsylvania
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Memphis, Tennessee
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Houston, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., McAllen, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., San Antonio, Texas
  - For information concerning this clinical site, please contact Nymox at 800-936-9669., Richmond, Virginia